CLINICAL TRIAL: NCT06395727
Title: Effect of Topical Airway Block on Hemodynamic Stability Post Induction of Anaesthesia in Cardiac Surgeries
Acronym: hemodynamics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R57/2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Surgery
Keywords: cardiac, airway block, lidocaine spray
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: Anaesthesia will be provided according to the hospital protocol in respect to preoperative investigations, fasting hours and intra-operative monitoring and drugs.
  All patients will be monitored by ECG, pulse oximeter and non-invasive blood pressure monitoring before receiving 2 mg midazolam for sedation before radial artery catheter insertion. After arterial catheter insertion, patients will be allocated to two groups, the first one (TBA group) will receive fentanyl traditional dose 3-5 mic/kg during induction. The second group will sit and receive lidocaine 2% nebulizer and then lidocaine 10 % oral application till achieving difficult swallowing. Then patient will lie, and induction will be done by fentanyl at a dose max 1 mic/kg. Then, both groups will receive general anaesthesia induction. Hemodynamic parameters will be recorded before induction, before intubation, 30 seconds, 1 minute and 2 minutes after intubation then every 5 minutes till skin incision.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- • Traditional balanced anaesthesia (control group) (Experimental): Analgesia will be offered by fentanyl 3-5 mic/kg in induction
  Interventions: Drug: Fentanyl
- • Airway topical anaesthesia (Experimental): Patient will be given lidocaine nebulizer (5 ml of lidocaine 2% with oxygen flow 8 l/m) after radial arterial catheter insertion that will be complemented by topical application of lidocaine spray 10 % not to exceed 200mg per dose on mouth with encouraging to move it in mouth then gargling with it before swallowing targeting reaching difficult swallowing.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Fentanyl — traditional fentanyl dose
  Arms: • Traditional balanced anaesthesia (control group)
Drug: Lidocain — lidocaine nebuliser and lidocaine spray targeting difficult swallowing
  Arms: • Airway topical anaesthesia

SUMMARY:
Opioids have always been the mainstay in management of patients during cardiac surgeries. Mega doses are often used to relieve stress of surgeries in highly labile patients with narrow hemodynamic threshold to keep the balance between oxygen demand and supply. Unfortunately, this is associated with hemodynamic instability and affect the fast-track pathway for extubation. Most of these doses are given in induction, so by blocking airway by non-invasive technique, this will help in the reduction in opioid doses and preventing risky hemodynamic instability during induction of anesthesia in these patients.

DETAILED DESCRIPTION:
Efficient handling of cardiac patients in cardiac surgeries is not an easy task. Patients are labile and more liable than others to hemodynamic changes in response to anaesthetic drugs and unfortunately, these changes are not well tolerated. (Choudhury A et al., 2017)

Any Hemodynamic change can have a great impact on the oxygen delivery - demand balance and lead to more damage. Every step is critical, but induction is the most challenging representing the peak of the dynamicity. Any change could happen, either tachycardia, hypertension, or arrhythmia in response to intubation or hypotension after induction or during period of minimal stimulus. (Soleimani A et al., 2017)

Although the concept of opioid based anaesthesia was the gold standard in cardiac surgeries for decades as opioids lack the negative inotropic effects, their usage was shifted from the mega doses of long acting opioids to titrating doses of short acting ones as fentanyl that became the primary in use.(Grant MC et al., 2023) Trying to control stress response to intubation by higher doses of opioids increase the liability for post induction hypotension which occurs in nearly one fourth to one third of patients receiving general anaesthesia. (Chen B et al., 2021)

The stress response to intubation could be inhibited by blocking the sensory pathway and hence the reflex response. Targeting the superior laryngeal nerve (SLN) that innervate the base of the tongue, epiglottis, piriform fossa, and vallecula together with trans tracheal topical anaesthesia will reduce the stress response to intubation. Fortunately, it's not essential to master anatomical landmarks and invasive techniques to block the sensory pathway as gradual topical spraying of local anaesthesia over the airway mucosal surfaces will lead to nearly equivalent effect in a simpler way. (Pignot G et al., 2022)

Lidocaine is one of the most commonly used local anaesthetics. It is generally safe and available in multiple dosage forms (topical, I.V., nebulizer and spray) and concentrations. It has been widely used for several indications in general anaesthesia starting from just cough suppression and reduction of sore throat to modulation of the stress response to intubation. (Mikawa K et al., 1997) Using lidocaine either topical or by nebulizer is a well-established method to anesthetise airway and can be used safely in cardiac surgeries. (Choudhury A et al., 2017) Also, lidocaine topical airway block showed significant effect on reducing QT changes in patients undergoing cardiac surgeries if applied before intubation. (Bilgi M et al.,2020)

Therefore, authors have hypothesised that air way block may help in reducing the doses of opioids needed to control the stress response of intubation and hence to better management of patient. This can be simply done by topical airway block with non-invasive techniques that are both safe and applicable for practice.

ELIGIBILITY:
Inclusion Criteria:

* • Undergoing elective cardiac surgery.

  * Age: above 18

Exclusion Criteria:

* • Pregnant or breast-feeding women

  * Emergency surgery
  * Anticipated difficult airway
  * Allergy to any of the drugs used in the study
  * Cannot cooperate to complete topical anaesthesia (with mental disorders or unable to communicate)
  * Use of a left ventricular assist device, IAB or ECMO prior to surgery
  * Presence of aortic dissection
  * EF<40 %
  * Severe mitral valve stenosis or severe aortic valve stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Hemodynamic instability | from induction to skin incision
  Hemodynamic instability before induction, before intubation and 30 seconds, 1 minute and 2 minutes after intubation then every 5 minutes till skin incision.

SECONDARY OUTCOMES:
Total doses of vasoactive drugs used | from induction to skin incision
  total dose of vaso active drugs used to support hemodynamics
Total doses of opioids used | through out the operation
  total dose of opioids used from induction to icu transferal

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Abdallah, Cairo
  - Abdallah Mahmoud Zaki Soudi, Cairo

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months